CLINICAL TRIAL: NCT02342457
Title: The Elactrophysiological Response of the Colon, in Normal Bowel, and Large Bowel Lacking Ganglia in Children With Suspected Hirschsprungs Disease.
Brief Title: Electrophysiological Activity of the Anorectum in Children Suspected of Hirschsprung Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Naftali Freud, Head of peadiatric surgery, Rabin Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0274-13-RMC
Record Dates: First submitted 2014-12-03; First posted 2015-01-21 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Hirschsprungs Disease
MeSH Terms: conditions — Hirschsprung Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Child suspected of Hirschsprung disease (Experimental): Children admitted for biopsy, so that Hirschsprungs desease may be ruled out or diagnosed, whom are planned for rectal biopsy, by clinical decision.
  Interventions: Device: Child suspected of Hirschsprung disease

INTERVENTIONS:
Device: Child suspected of Hirschsprung disease — Children admitted for rectal biopsy, due to chronic constipation and suspected of Hirschsprungs disease, will undergo electrophysiological reading from the rectal inner wall, at thechosen site for biopsy before biopsy is performed. Histopathology and readings will be analyzed for corelation
  Other Names: Electrophysiological study of the rectum in children

SUMMARY:
Children with chronic constipation, suspected of having hirschsprungs disease, who are admitted for rectal biopsy will be included in the study. During the procedure, electrophysiological reading from the site chosen for biopsy will be done. Correlation between electrophysiological data and histopathology will be analyzed.

DETAILED DESCRIPTION:
Hirschsprungs disease is found in 1:5000 newborns, the disease is caused by aganglionosis of the colon, leading to severe constipation and possible bowel obstruction. The diagnosis is based on leveling biopsies taken from the rectum and colon. Treatment is supportive if complications had arisen, and surgical for definitive correction of the pathophysiological condition which is the cause of the disease. Currently, clinicians rely on histopathology, for diagnosing the disease, and planning surgical correction. The main goal of Surgical treatment will be the creation of a continuous patent and innervated bowel, in which effective propulsive peristalsis is taking place. This is achieved by resection of aganglionic colon, and anastomosis of normal colon with normal ganglia, to anus. Today surgeons await histopathology report for the diagnosis of Hirschsprungs disease, and frozen section biopsies taken when in surgery to ascertain the level of ganglionated bowel.

In this study the investigators aim to correlate electrophysiological reading, from colon suspected of Hirschsprungs disease. If correlation is found, or a specific pattern which is diagnostic of the disease may be found, the electrophysiological study may offer a new way of diagnosing the disease, which is not invasive and allows prompt diagnosis in contrast to histopathology which is time consuming. A reliable electrophysiological study for Hirschsprungs disease may be helpful in early and correct diagnosis, with a noninvasive procedure as compared to a biopsy of the colonic wall. Children with chronic constipation, suspected of having hirschsprungs disease, who are admitted for rectal biopsy will be included in the study. During the procedure, electrophysiological reading from the site chosen for biopsy will be done. Correlation between electrophysiological data and histopathology will be analyzed. The actual reading will be carried out by a custom made electrode by GAELTEC DEVICES LTD : DUNVEGAN : ISLE OF SKYE : SCOTLAND.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted for rectal biopsy, by clinical decision, so that Hirschsprungs disease may be diagnosed or ruled out

Exclusion Criteria:

None

-

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-03; Primary Completion 2017-03 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Characteristic electrophysiologic curve for aganglionated bowel | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Freud, MD, Principal Investigator — Schneider medical center of Israel

REFERENCES:
- [Background] Marin AM, Rivarola A, Garcia H. Electromyography of the rectum and colon in Hirschsprung's disease. J Pediatr Surg. 1976 Aug;11(4):547-552. doi: 10.1016/s0022-3468(76)80010-3. PMID 787484